CLINICAL TRIAL: NCT00673881
Title: ABT-335 (Choline Fenofibrate)Reverse Cholesterol Transport (RCT) Study
Brief Title: ABT-335 (Choline Fenofibrate) Reverse Cholesterol Transport (RCT) Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radiant Research (Other)
Responsible Party: Michael H. Davidson,MD, FACC, Radiant Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-335-001
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Results first posted 2011-04-20 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-03

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abt-335 (Experimental): ABT-335 (choline fenofibrate)
  Interventions: Drug: choline fenofibrate

INTERVENTIONS:
Drug: choline fenofibrate — 135 mg choline fenofibrate daily(oral, capsule)
  Other Names: ABT-335

SUMMARY:
The objectives of the study are:

1. To evaluate the effect of ABT-335 (choline fenofibrate) on several parameters of RCT (reverse cholesterol transport) in men and post-menopausal women diagnosed with dyslipidemia (i.e., low high-density lipoprotein [HDL] cholesterol levels and elevated triglyceride [TG] concentrations).
2. To evaluate longitudinal changes in several parameters of RCT in subjects with low HDL.
3. To obtain pilot data for power calculations for subsequent comparative study.

DETAILED DESCRIPTION:
This trial assesses the effects of ABT-335 on RCT as measured by cholesterol efflux or rate of appearance of cholesterol (Ra in mg/kg/hr), cholesterol excretion (%/day), RCT efflux (mg/kg/day) and de novo cholesterol synthesis (%) during a baseline period (7 days) and during a treatment period (94 days).

The goal of using RCT to reverse atherosclerosis is to increase the rate of cholesterol export or "efflux" from the tissues and plaques. An increase in this cholesterol efflux rate should shrink arterial plaques by decreasing their static accumulation of cholesterol. While some currently marketed drugs have a positive impact on RCT by increasing the rate of cholesterol excretion from the body, no drug has yet been approved to increase the rate of cholesterol efflux from the tissues

ELIGIBILITY:
Inclusion Criteria:

1. Male, non-smoker, 21 - 75 years of age inclusive.
2. Female, non-smoker, 40 - 75 years of age inclusive.
3. Post-menopausal women, as defined by lack of menses for at least 2 years and age > 55, OR history of documented bilateral surgical oophorectomy, confirmed with an elevated follicle-stimulating hormone (FSH) at screening.
4. HDL concentration (≤ 50 mg/dl women, ≤ 40mg/dl men)
5. TG concentration 150-500 mg/dl, inclusive
6. Ability to give informed consent

Exclusion Criteria:

1. Subject has history of diabetes mellitus, active hepatitis, gall bladder disease, gastric bypass surgery, or clinically significant abnormalities on screening (prestudy) physical examination or laboratory tests.
2. Screening laboratory tests with hematocrit <30%, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) > 2X upper limit of normal, abnormal thyroid-stimulating hormone (TSH), fasting glucose ≥126 mg/dl.
3. Renal impairment with creatinine clearance < 80 ml/min.
4. Treatment within the last 6 months with drugs known to alter lipid metabolism including beta blockers, thiazide diuretics, bile acid resins, ezetimibe, fibrates, niacin, and fish oils (see Appendix 1). Washout of fibrates is not permitted.
5. Treatment with drugs known to interact with ABT-335, e.g., warfarin (see Appendix 1).
6. Treatment with HMG CoA reductase inhibitors (statins) within the past 4 weeks (see Appendix 1).
7. History of allergy to egg or soy products.
8. History of coronary heart disease (CHD), stroke or revascularization procedure in the six months prior to Visit 1.
9. Current or recent history (past 12 months) of drug abuse or alcohol abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor).
10. Participation in another clinical trial or exposure to any investigational agent within 30 days before visit 1.
11. Individual has a condition the Principal Investigator believes would interfere with his/her ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the subject at undue risk.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Davidson, MD,FACC, Principal Investigator — Radiant Research
Locations (1):
- Radiant Research, 515 N State St, #2700, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ABT 335: choline fenofibrate, 135 mg/day,orally, 12 weeks
Period: Overall Study
Arm/Group | ABT 335
Started | 25
Completed | 24
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | ABT 335
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 25
Total cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] — Mean of fasting (> 12 hours) total cholesterol measured at screening, Day 0, 1PM and Day 1, 1AM (Visit 1),Day 10 (Visit 4);23 values, per protocol population
  mg/dL | 221 (45)
Triglycerides (TG) [Mean (Standard Deviation); unit: mg/dL] — Mean fasting (> 12 hours) triglycerides measured at screening, Day 0, 1PM and Day 1, 1AM (Visit 1), Day 10 (Visit 4);23 values, per protocol population
  mg/dL | 241 (122)
High Density Lipoprotein Cholesterol (HDL) [Mean (Standard Deviation); unit: mg/dL] — Mean fasting (> 12 hours) HDL cholesterol measured at screening, Day 0, 1PM and Day 1, 1AM (Visit 1), Day 10 (Visit 4); 23 values, per protocol population
  mg/dL | 34 (8.2)
Low density lipoprotein cholesterol (LDL) [Mean (Standard Deviation); unit: mg/dL] — Mean fasting (> 12 hours) LDL cholesterol measured at screening, Day 0, 1PM and Day 1, 1AM (Visit 1), Day 10 (Visit 4); 23 values, per protocol population
  mg/dL | 144 (40)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Calculated Low Density Lipoprotein Cholesterol
Description: Mean change in calculated LDL, baseline (average Day 0, 1 10) to end-of-treatment (12 weeks treatment,average Day 95)
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ABT 335
Number analyzed (Participants) | 23
mg/dL | -22.7 (34.2)
Statistical Analysis 1: Comparison: ABT 335; Test type: Superiority or Other; p = 0.0042, t-test, 2 sided

2. Primary Outcome: Mean Change in Plasma Triglycerides
Description: Change in plasma triglyceride, baseline (average Day 0, 1 10) to end-of-treatment (12 weeks treatment,Day 95)
Time Frame: baseline to 12 weeks
Population: per protocol
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ABT 335
Number analyzed (Participants) | 23
mg/dL | -138.0 (150.5)
Statistical Analysis 1: Comparison: ABT 335; Comparison baseline to end-of-treatment; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided

3. Primary Outcome: Mean Change in High Density Lipoprotein Cholesterol
Description: Mean change in plasma high density plasma lipoprotein cholesterol (HDL-C)baseline (average Day 0, 1 10) to end-of-treatment (12 weeks treatment,Day 95)
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ABT 335
Number analyzed (Participants) | 23
mg/dL | -1.6 (6.0)
Statistical Analysis 1: Comparison: ABT 335; Comparison from baseline to end-of-treatment; Test type: Superiority or Other; p = NS, t-test, 2 sided

4. Secondary Outcome: Plasma Cholesterol Efflux
Description: Change in efflux rate from baseline to end-of-treatment. The efflux rate of cholesterol from peripheral tissues into the plasma was measured as mg/kg/hr. An IV infusion of [13C2] cholesterol mixed in 10% Intralipid® or Liposyn® and 10 % ethanol was given piggy-backed into normal saline over 24 hours. This was used to determine rate of appearance (Ra) cholesterol, measured by dilution of infused [13C2] cholesterol during the plateau phase of plasma enrichment (approximately the last 4 hours of the infusion), as well as to provide the plasma cholesterol traced into biliary sterols.
Time Frame: 12 weeks
Reporting Status: Not Posted
Measure: Mean (Full Range); unit: mg/kg/hr

5. Secondary Outcome: Change in Plasma Cholesterol Ester Fractional Catabolic Rate (FCR)
Description: Change in FCR from baseline to end-of-treatment (12 weeks)
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted
Measure: Number; unit: mg/kg/day

6. Secondary Outcome: Percent Change in de Novo Cholesterol Synthesis
Description: Plasma DNC was measured three times from blood draws on the 3 visits in the 10 day period following the isotope infusion at baseline and again at end-of-treatment at 12 weeks, and expressed in percent. Change from baseline to end-of-treatment expressed as percent.
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted
Measure: Number; unit: change, percent

7. Secondary Outcome: Change in Neutral Sterol Excretion
Description: The excretion rate of fecal neutral and acidic sterols was measured as mg/day, for each individual three times during the 10 day period following the isotope infusions at baseline and end-of-treatment.
Time Frame: baseline to 12 weeks
Reporting Status: Not Posted
Measure: Number; unit: Change, mg/day

8. Secondary Outcome: Change in Bile Acid Excretion
Description: Change in bile acid excretion from baseline to end-of-treatment
Time Frame: Baseline to 12 weeks
Reporting Status: Not Posted
Measure: Number; unit: percent change

9. Secondary Outcome: Neutral Sterol Endogenous Excretion
Description: Change in neutral sterol endogenous excretion from baseline to end-of-treatment
Time Frame: 12 weeks
Reporting Status: Not Posted
Measure: Number; unit: percent

10. Secondary Outcome: Endogenous Bile Acid Excretion
Description: Change in endogenous bile acid excretion from baseline to end-of-treatment
Time Frame: 12 weeks
Reporting Status: Not Posted
Measure: Number; unit: percent

11. Primary Outcome: Total Cholesterol
Description: Mean Change in total cholesterol from baseline to End-of-treatment (Day 95)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ABT 335
Number analyzed (Participants) | 23
mg/dL | -54.0 (34.4)
Statistical Analysis 1: Comparison: ABT 335; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: All adverse events occurring during the study are reported - the study included a treatment period, with pre-study baseline and post-study end-of-treatment procedures.
Arm/Group | ABT 335
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 14/25
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT 335 (N=25)
diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 2
back pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 2
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes